CLINICAL TRIAL: NCT05988359
Title: Assessment of Aerosol Quantity Generated During Caries Treat-ment With Er:YAG Laser. A Randomized Clinical Trial.
Brief Title: Quantitative Evaluation of Aerosols Produced in the Dental Office
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jacek Matys, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU4
Record Dates: First submitted 2023-06-28; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Aerosol Disease; Caries,Dental
Keywords: laser; Er:YAG; disinfection; bacteria; high-volume evacuator
MeSH Terms: conditions — Dental Caries | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental turbine (Active Comparator): In the first group, G1 (n=30) a conventional high-volume evacuator (Monoart® Euronda, Vicenza, Italy) was used to remove aerosols during caries treatment by a dental turbine.
  Interventions: Procedure: Caries treatment with a dental turbine
- Laser (Experimental): In the second G2 (test, n=30) group, a conventional high-volume evacuator (Monoart® Euronda, Vicenza, Italy) was used to remove aerosols during caries treatment by an Er:YAG laser.
  Interventions: Procedure: Caries treatment with Er:YAG laser

INTERVENTIONS:
Procedure: Caries treatment with a dental turbine — G1 (n=30) conventional high-volume evacuator (Monoart® Euronda, Vicenza, Italy) was used to remove aerosols during caries treatment.
  Arms: Dental turbine
Procedure: Caries treatment with Er:YAG laser — G2 (test, n=30) group, a conventional high-volume evacuator (Monoart® Euronda, Vicenza, Italy) was used to remove aerosols during caries treatment.
  Arms: Laser

SUMMARY:
Background: Maintaining biosafety in dental practice requires an efficient elimination of aerosols produced during dental treatment. The objective of this research was to assess the quantity of aerosols and aerobic bacteria present in the air during the treatment of caries. Methods: This study was divided into two groups based on the caries treatment method involving 60 patients with 60 m olar teeth (n=60) in the mandible. Group 1 (n=30) received a conventional dental turbine W&H Synea TA-98LC (W&H, Bürmoos, Austria), while Group 2 (n=30) received an Er:YAG laser (LightWalker, Fotona, Slovenia). Measurements of aerosol particles between 0.3 - 10.0 μm near the operator's mouth were taken using the PC200 laser particle counter (Trotec GmbH, Schwerin, Germany). The number of aerobic bacteria in the air was determined using 60 micro-biological plates with a microbiological medium (Columbia Agar with 5% Sheep Blood) and the sedimentation method. A control group G3 was established to measure the initial aero-sol level and the initial total number of bacteria CFUs (colony-forming units) before each treatment.

ELIGIBILITY:
Inclusion Criteria:

- The subjects were chosen for the study under the subsequent inclusion criteria: occurrence of medium or profound caries on Black class I, ICDAS 3,4

Exclusion Criteria:

* Patients with systematic diseases that can influence the treatment of periodontitis
* Patients under or took antibiotics 2 months.
* Patients under or took immunosuppressors the last 6 months.
* Pregnant or lactating woman.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Aerosols measurment | immediately before the procedure
  The aerosols were measured with a PM200 detector counter (Trotec GmbH, Schwerin, Germany).
Aerosols measurment | immediately after the procedure
  The aerosols were measured with a PM200 detector counter (Trotec GmbH, Schwerin, Germany).

SECONDARY OUTCOMES:
Bacteriological study | 60 miniutes before the procedure
  The total number of aerobic bacteria in the air of the dental office was carried out by the Koch sedimentation method. The study used 60 Petri dishes with a microbiological medium (Columbia Agar with 5% Sheep Blood) to check the number of aerobic bacteria. Twenty plates were opened 60 minutes before the study (control group, n=20) and closed before the start of caries treatment. Next, forty plates were opened at the start of car-ies treatment with additional using a conventional evacuator (n=20) or a new evacuator (n=20) and closed 60 minutes after the treatment.
Bacteriological study | immediately before the procedure
  The total number of aerobic bacteria in the air of the dental office was carried out by the Koch sedimentation method. The study used 60 Petri dishes with a microbiological medium (Columbia Agar with 5% Sheep Blood) to check the number of aerobic bacteria. Twenty plates were opened 60 minutes before the study (control group, n=20) and closed before the start of caries treatment. Next, forty plates were opened at the start of car-ies treatment with additional using a conventional evacuator (n=20) or a new evacuator (n=20) and closed 60 minutes after the treatment.
Bacteriological study | immediately after the procedure
  The total number of aerobic bacteria in the air of the dental office was carried out by the Koch sedimentation method. The study used 60 Petri dishes with a microbiological medium (Columbia Agar with 5% Sheep Blood) to check the number of aerobic bacteria. Twenty plates were opened 60 minutes before the study (control group, n=20) and closed before the start of caries treatment. Next, forty plates were opened at the start of car-ies treatment with additional using a conventional evacuator (n=20) or a new evacuator (n=20) and closed 60 minutes after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Surgery Department, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No